CLINICAL TRIAL: NCT01843673
Title: Image-Guided Adaptive Radiotherapy for Head And Neck Cancer: Patient Image Acquisition
Brief Title: Image-Guided Adaptive Radiotherapy for in Detecting Tumors During Treatment in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MCC-11639; NCI-2013-00846 (Registry Identifier: NCI); HM11639 (Other: Virginia Commonwealth University IRB)
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-05

CONDITIONS: Head and Neck Cancer
Keywords: Lip, Oral Cavity and Pharynx; Larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphoid Interstitial Pneumonia; Laryngeal Diseases | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- in-room imaging systems (Experimental): Patients undergo FBCT once before treatment and once weekly for a total of 6-7 scans, dual CBCT up to 5 times weekly for a total of 33-35 scans, 2-D x-ray with Varian kV OBI 5 times weekly for a total of 33-35 scans, 2-D x-ray with Brain Lab ExacTrac 5 times weekly for a total of 33-35 scans, 2-D x-ray with Varian MV OBI once weekly for a total of 6-7 scans, and EPID imaging up to 5 times weekly for a total of 33-35 scans while undergoing IGART.
  Interventions: Procedure: computed tomography; Procedure: cone-beam computed tomography; Procedure: radiography; Procedure: electronic portal imaging; Radiation: image-guided adaptive radiation therapy

INTERVENTIONS:
Procedure: computed tomography — Undergo FBCT
  Other Names: tomography, computed
Procedure: cone-beam computed tomography — Undergo dual CBCT
Procedure: radiography — Undergo 2-D x-ray with Varian kV OBI
  Other Names: Conventional X-Ray, Diagnostic Radiology, Medical Imaging, X-Ray, X-Ray Imaging
Procedure: radiography — Undergo 2-D x-ray with Brain Lab ExacTrac
  Other Names: Conventional X-Ray, Diagnostic Radiology, Medical Imaging, X-Ray, X-Ray Imaging
Procedure: radiography — Undergo 2-D x-ray with Varian MV OBI
  Other Names: Conventional X-Ray, Diagnostic Radiology, Medical Imaging, X-Ray, X-Ray Imaging
Procedure: electronic portal imaging — Undergo EPID imaging
  Other Names: EPI
Radiation: image-guided adaptive radiation therapy — Undergo IGART
  Other Names: IGART, image-guided adaptive radiotherapy

SUMMARY:
This clinical trial studies image-guided adaptive radiotherapy in detecting tumors during treatment in patients with head and neck cancer. Image-guided adaptive radiotherapy uses high quality imaging technology to detect the tumor and normal organs during treatment. It is not yet known which imaging technique provides the best image for guidance during treatment with radiation therapy. Comparing results of imaging procedures done before, during, and after radiotherapy may help doctors plan the best treatment.

DETAILED DESCRIPTION:
I. To conduct a clinical imaging study utilizing three novel in-room imaging systems: Oblique Brainlab ExacTrac images, Orthogonal Varian kilovoltage (kV) On-board Imaging (OBI) image, and Varian cone-beam computed tomography (CBCT) imaging to assess their performance in reducing inter- and intrafractional setup errors, relative to weekly megavoltage (MV) electronic portal imaging device (EPID) images, using both bony landmarks and soft tissue changes for head and neck cancer (HNC) patients undergoing external beam radiation therapy (RT).

II. To assess the accuracy of CBCT imaging for measuring systematic soft tissue changes in the head and neck (HN) area relative to conventional high resolution contrast enhanced fan-beam computed tomography (CT) (FBCT) as a standard.

III. To assess the systematic and random soft tissue motion errors using daily CBCT imaging relative to bony-landmark alignment to evaluate the benefit of soft tissue imaging during radiotherapy.

IV. To quantify soft tissue changes during an entire course of radiotherapy (e.g. tumor shrinkage) using daily CBCT imaging.

V. To determine the feasibility of using measured set up and soft-tissue motion uncertainties in conjunction with volume changes observed on serial CBCT images, for offline adaptive replanning of HNC patients using available planning tools.

VI. To quantify the benefits of adaptive image-guided radiotherapy (IGRT) in HN patients in terms of target coverage and normal tissue avoidance.

VII. To determine the feasibility of mounting a phase I/II trial to assess the clinical benefits of image-guided adaptive radiotherapy (IGART) in terms of acute and late toxicities and tumor control.

VIII. To build a HNC patient database for future validation of IGART processes using deformable image registration and Virtual Clinical Trials (VCTs).

OUTLINE:

Patients undergo FBCT once before treatment and once weekly for a total of 6-7 scans, dual CBCT up to 5 times weekly for a total of 33-35 scans, 2-dimensional (2-D) x-ray with Varian kV OBI 5 times weekly for a total of 33-35 scans, 2-D x-ray with Brain Lab ExacTrac 5 times weekly for a total of 33-35 scans, 2-D x-ray with Varian MV OBI once weekly for a total of 6-7 scans, and EPID imaging up to 5 times weekly for a total of 33-35 scans while undergoing IGART.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of head and neck malignancy
* Patients who will be treated with definitive radiation therapy or concurrent chemoradiation therapy
* Gross tumor volume (GTV) must be visible on CT
* All patients must be informed of the investigational nature of this study and must give written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Pregnant or nursing women may not participate; women of reproductive potential must be offered a pre-treatment pregnancy test and informed of the need to practice an effective contraceptive method
* Prior treatment with radiation therapy to the head and neck
* Serum creatinine > 1.5 and/or
* Blood urea nitrogen [BUN] > 25
* Treatment with any prior chemotherapy or surgery (excluding diagnostic biopsy) for this malignancy
* Patients with known syndromes expected to alter radiosensitivity (e.g. ataxia-telangiectasia, scleroderma, lupus, human immunodeficiency virus [HIV]/acquired immunodeficiency deficiency syndrome [AIDS]) may not participate

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Evans, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Massey Cancer Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (Imaging Technology): Patients undergo FBCT once before treatment and once weekly for a total of 6-7 scans, dual CBCT up to 5 times weekly for a total of 33-35 scans, 2-D x-ray with Varian kV OBI 5 times weekly for a total of 33-35 scans, 2-D x-ray with Brain Lab ExacTrac 5 times weekly for a total of 33-35 scans, 2-D x-ray with Varian MV OBI once weekly for a total of 6-7 scans, and EPID imaging up to 5 times weekly for a total of 33-35 scans while undergoing IGART.
  computed tomography: Undergo FBCT cone-beam computed tomography: Undergo dual CBCT radiography: Undergo 2-D x-ray with Varian kV OBI radiography: Undergo 2-D x-ray with Brain Lab ExacTrac radiography: Undergo 2-D x-ray with Varian MV OBI electronic portal imaging: Undergo EPID imaging image-guided adaptive radiation therapy: Undergo IGART
Period: Overall Study
Arm/Group | Diagnostic (Imaging Technology)
Started | 16
Completed | 10
Not Completed | 6
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Imaging Technology)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Differences of Calculated Set up Errors of 2 mm Between the Different Imaging Technologies
Description: The automated patient setup procedure varies between 'OBI', 'CBCT' or 'Exactrac' imaging technologies. Each procedure gives two shifts: 'vertical' and 'lateral'. In the absence of a gold standard, our goal is to compare the shifts recommended by each pair of automated patient setup procedures. Average and Std deviation of vertical and lateral motion from the three systems were computed. P value, 1.00, refers to the test of difference of each system with OBI being more than 2 mm. Pairwise comparison for each direction between each pair of technologies were done using a t test to check if the difference in the recommended shift is more than 2 mm. The reported mean value represents the shift from planned treatment position averaged over all daily treatment setups. A negative mean vertical value indicates the patient was consistently set up posterior to plan; a negative mean lateral value indicates a set up consistently right of plan.
Time Frame: up to 7 weeks
Population: Ten evaluable head and neck patients treated with external beam radiation therapy received 19 to 32 fractions with all three imaging techniques. The mean daily shift of these 19 to 32 fractions were recorded for each technique. Statistical significance is determined based on 5% level of significance.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Orthogonal Varian kV OBI Image: Patients are first set up for treatment with surface fiducial marks and followed by an automated image guided alignment procedure to achieve better alignment with the planning image. The automated procedure OBI gives two shifts: vertical and lateral. In the absence of a gold standard, our goal is to compare the vertical and lateral shifts recommended by each pair of automated procedures.
- Varian CBCT (Cone Beam CT) Imaging: Patients are first set up for treatment with surface fiducial marks and followed by an automated image guided alignment procedure to achieve better alignment with the planning image. The automated procedure CBCT gives two shifts: vertical and lateral. In the absence of a gold standard, our goal is to compare the vertical and lateral shifts recommended by each pair of automated procedures.
- Oblique Brainlab ExacTrac Images: Patients are first set up for treatment with surface fiducial marks and followed by an automated image guided alignment procedure to achieve better alignment with the planning image. The automated procedure ExacTrac gives two shifts: vertical and lateral. In the absence of a gold standard, our goal is to compare the vertical and lateral shifts recommended by each pair of automated procedures.
Arm/Group | Orthogonal Varian kV OBI Image | Varian CBCT (Cone Beam CT) Imaging | Oblique Brainlab ExacTrac Images
Number analyzed (Participants) | 10 | 10 | 10
mm
  Vertical shift | -1.2 (3.1) | -0.8 (3.4) | -1.8 (3.2)
  Lateral shift | -1.5 (3.3) | -1.1 (3.3) | 1.3 (3.9)
Statistical Analysis 1: Comparison: Orthogonal Varian kV OBI Image vs Varian CBCT (Cone Beam CT) Imaging; Pairwise comparison for each direction between each pair of technologies were done using a t test to check if the difference in the recommended shift is more than 2 mm. Clinical significance is based on a 2 mm difference. Statistical significance is determined based on 5% level of significance; Test type: Non-Inferiority or Equivalence — Statistical significance testing at 5% level of significance, p-value being larger than 0.05 . The p-values for pairwise comparison; p = 1.00, t-test, 2 sided — Statistical significance testing at 5% level of significance, p-value being larger than 0.05. The p-values for pairwise comparison lateral and vertical, for OBI and CBCT was 1.00
Statistical Analysis 2: Comparison: Orthogonal Varian kV OBI Image vs Oblique Brainlab ExacTrac Images; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Statistical significance testing at 5% level of significance, p-value being larger than 0.05. Those are the p-values for pairwise comparison; p = 1.00, t-test, 2 sided — Statistical significance testing at 5% level of significance, p-value being larger than 0.05. The p-values for pairwise comparison lateral and vertical, for OBI and ExacTrac was 1.00

2. Primary Outcome: Dose Variation Between the Different Imaging Technologies for Normal Tissue Structures of 10%
Time Frame: Up to 7 weeks
Population: No data analyzed due to staff leaving primary institution.
Arm/Group | Orthogonal Varian kV OBI Image | Varian CBCT (Cone Beam CT) Imaging | Oblique Brainlab ExacTrac Images
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Greater Than or Equal to 5% Variation of Normal Tissue Toxicity
Time Frame: Up to 7 weeks
Population: No data analyzed due to staff leaving primary institution.
Arm/Group | Orthogonal Varian kV OBI Image | Varian CBCT (Cone Beam CT) Imaging | Oblique Brainlab ExacTrac Images
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event Reporting were collected up to 7 weeks while the patient was undergoing the course of radiation therapy. No adverse events occurred due to additional xray imaging from this study.
Arm/Group | Diagnostic (Imaging Technology)
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 7/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Imaging Technology) (N=16)
SEPSIS-ASSOCIATED ORGAN DYSFUNCTION (Infections and infestations) | 1 (1) — Death not associated with CTCAE term - Sudden death. Cause of Death, SEPSIS-ASSOCIATED ORGAN DYSFUNCTION
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Imaging Technology) (N=16)
Below normal Glomerular filtration rate (GFR) (Blood and lymphatic system disorders) | 2 (2) — Metabolic/Laboratory, Glomerular filtration rate grade 1 and grade 2
Elevated Creatinine (Blood and lymphatic system disorders) | 6 (7) — 3 events grade 1 and 4 events grade 2.
Elevated Blood Urea Nitrogen (BUN) (Blood and lymphatic system disorders) | 3 (3) — Metabolic/Laboratory - Other (Specify, __)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes